CLINICAL TRIAL: NCT03557112
Title: Prospective, Multicenter, and Nonrandomized Phase II Clinical Study on the Treatment of Locally Advanced NPC By Comparing TPF Induction Chemotherapy Combined With Nimotuzumab Concurrent Radiotherapy and Cisplatin Concurrent Radio-chemotherapy
Brief Title: By Comparing TPF Induction Chemotherapy Combined With Nimotuzumab Concurrent Radiotherapy and Cisplatin Concurrent Radio-chemotherapy for Locally Advanced NPC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guiyang Medical University (Other)
Responsible Party: Principal Investigator, Feng Jing, Head and neck cancer director, chief researcher, clinical professor, Guiyang Medical University
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20180604
Record Dates: First submitted 2018-06-04; First posted 2018-06-14 (Actual); Last update posted 2018-11-02 (Actual); Status verified 2018-06

CONDITIONS: Nasopharyngeal Carcinoma
Keywords: Locally Advanced Nasopharyngeal Carcinoma; nimotuzumab; chemoradiotherapy; cisplatin
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — nimotuzumab; Cisplatin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- the treatment group (Experimental): TPF regimen induction chemotherapy combined with nimotuzumab concurrent radiotherapy concurrent chemoradiotherapy
  Interventions: Drug: Nimotuzumab
- the control group (Active Comparator): TPF regimen induction chemotherapy combined with cisplatin concurrent radiotherapy concurrent chemoradiotherapy
  Interventions: Drug: Cisplatin

INTERVENTIONS:
Drug: Nimotuzumab — TPF Regimen Induction Chemotherapy combined with nimotuzumab concurrent radiotherapy concurrent chemoradiotherapy
  Other Names: Nimotuzumab lnjection
  Arms: the treatment group
Drug: Cisplatin — TPF Regimen Induction Chemotherapy combined with cisplatin concurrent radiotherapy concurrent chemoradiotherapy
  Other Names: cis-DDP; cis-Diammineplatinum(II) dichloride
  Arms: the control group

SUMMARY:
This study is aimed to investigate the short-term efficacy and toxicities of local advanced nasopharyngeal carcinoma (NPC) treated with TPF regimen induction chemotherapy combined with nimotuzumab concurrent radiotherapy and cisplatin concurrent chemoradiotherapy.

DETAILED DESCRIPTION:
TPF program is currently the local advanced nasopharyngeal carcinoma commonly used inducing chemotherapy, cisplatin is the preferred drug for the same period chemotherapy, however, due to heavier gastrointestinal reactions caused by cisplatin， direct damage to renal parenchymal and other adverse reactions often lead to anti-tumor therapy can not be smooth Carried out, resulting in treatment failure, thus affecting the survival of patients.In this study, Phase II clinical trials were performed. Patients with locally advanced local advanced nasopharyngeal carcinoma were nonrandomly divided into experimental group and control group.The trial group was treated with TPF regimen induction chemotherapy combined with nimotuzumab concurrent radiotherapy and chemotherapy. The control group was treated with TPF regimen induction chemotherapy combined with Cisplatin concurrent radiotherapy and chemotherapy.observed and compared the efficacy and toxicity of the two treatment to assess its safety and patient tolerance.

ELIGIBILITY:
Inclusion Criteria:

1. The pathological type is non-keratinizing cancer (according to the World Health Organization, WHO pathological classification).
2. The stage is graded by TxNxM0 (according to the eighth edition of the AJCC staging standard).
3. Age: Between 18 to 70.
4. EGFR, which is performed by biopsy immunohistochemical examination, shows positive.
5. Functional Status: Karnofsky Scale (KPS) > 70.
6. Normal Bone Marrow Function: White blood cell count > 4×109/L, hemoglobin >90g/L, and platelet count >100×109/L.
7. Normal Liver Function: Alanine Tminotransferase (ALT), Aspartate Aminotransferase (AST) < 1.5 times the upper limit of normal (ULN), while alkaline phosphatase (ALP) < 2.5 x ULN and bilirubin < ULN.
8. Normal Renal Function: creatinine clearance > 60 ml/min.
9. The patient must be informed of the basic content of the study and sign an informed consent.

Exclusion Criteria:

1. Patients with a prior history of malignant tumors, except well-treated basal cell carcinoma or squamous-cell carcinoma, and cervical carcinoma in situ.
2. Women during pregnancy or breastfeeding (for women of child-bearing age, pregnancy test should be considered; effective contraception should be emphasized during treatment).
3. Patients received radiotherapy, chemotherapy, and immunological targeted therapies (non-melanoma skin cancers with previous lesions outside the target of radiotherapy are excluded).
4. Patients received treatments for primary lesions and metastatic cervical lesions (except diagnostic treatment).
5. Patients with other serious diseases which may bring greater risk or affect the compliance of the trial. For example: unstable heart disease requiring treatment, kidney disease, chronic hepatitis, uncontrolled diabetes (fasting blood glucose >1.5 x ULN), and mental illness.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2018-06-01 (Actual); Primary Completion 2021-06-01 (Estimated); Study Completion 2021-12-01 (Estimated)

PRIMARY OUTCOMES:
National Cancer Institute CTCAE v4.0 | 1 year
  Acute toxicity of radiotherapy and chemotherapy

SECONDARY OUTCOMES:
evaluation of immediate efficacy overall survival overall survival overall survival overall survival overall survival overall survival | 1 year
  Evaluation of efficacy by RESIST1.1 standard
overall survival | 5 years
  Evaluate the Overall survival after Concurrent chemo-radiotherapy by RECIST
locoregional failure-free survival | 5 years
  Evaluate the Overall survival after Concurrent chemo-radiotherapy by RECIST
progression-free survival | 5 years
  Evaluate the Overall survival after Concurrent chemo-radiotherapy by RECIST

CONTACTS AND LOCATIONS:
Overall Officials: Feng Jin, Bachelor, Study Chair — Guizhou Provincial Cancer Hospital
Locations (1):
- Cancer Hospital of Guizhou Medical University, Guiyang, Guizhou, China

IPD SHARING:
Plan to Share IPD: No